CLINICAL TRIAL: NCT00131872
Title: Clinical Study Comparing Expedial and ePTFE Vascular Access Grafts
Brief Title: Study to Evaluate the Performance and Safety of Expedial and Compare it to Expanded Polytetrafluoroethylene (ePTFE) Vascular Access Grafts
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: LeMaitre Vascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00168
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2006-11

CONDITIONS: End Stage Renal Disease
Keywords: vascular access graft; hemodialysis; dialysis; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Device: Expedial Vascular Access Graft

SUMMARY:
The purpose of this study is to establish the substantial equivalence of Expedial and ePTFE grafts for effectiveness in maintaining primary or assisted primary patency.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic renal failure and requires vascular access for hemodialysis
* Patient has given informed consent to participate in the trial and is willing to comply with the study protocol
* Patient is male or female, 18 years of age or older
* The vascular access graft can be placed in the upper extremity (forearm, including across the elbow, or upper arm)
* Patient is undergoing or will undergo hemodialysis at a hospital or hemodialysis center
* Patient has a vein 4 mm or larger to which the graft can be anastomosed

Exclusion Criteria:

* Patient is unable to comply with the study follow-up
* Patient has a known sensitivity to polyurethane or porcine heparin
* Patient has a previous vascular access graft implanted and it is not possible to place the study graft proximal to the existing device and no other sites are available
* Patient has an immunodeficiency syndrome
* Patient has a prior history of bacterial infection within 8 weeks of implantation of graft
* Patient has a severe coagulation disorder
* Patient has an elevated platelet count of greater than 1 million
* Patient has a history of heparin-induced thrombocytopenia syndrome (HIT)
* Patient is pregnant
* Patient has a fever greater than 100 degrees Fahrenheit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2004-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Primary or assisted primary patency at 1 year

SECONDARY OUTCOMES:
Secondary patency
Overall adverse event rate
Time to first access
Time to hemostasis following needle withdrawal after dialysis

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Vascular and General Surgery, Miami, Florida
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - Vascular Surgery, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - General Surgery, Bamberg, South Carolina
  - South Carolina Associates for Cardiac and Vascular Disease; Greenville Hospital System, Greenville, South Carolina
  - Peripheral Vascular Associates, San Antonio, Texas